CLINICAL TRIAL: NCT01213238
Title: A Phase I Clinical Trial of Hepatic Arterial Infusion of Oxaliplatin, Oral Capecitabine, With or Without Systemic Bevacizumab for Patients With Advanced Cancer Metastatic to the Liver
Brief Title: Hepatic Arterial Infusion Oxaliplatin, Capecitabine With or Without Bevacizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0413; NCI-2012-01901 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Advanced Cancers
Keywords: Liver metastasis; hepatic arterial infusion; HAI; Eloxatin; Xeloda; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Oxaliplatin; Capecitabine; Bevacizumab
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxaliplatin + Capecitabine + Bevacizumab (Experimental): Oxaliplatin 140 mg/m2 by Hepatic Arterial Catheter (HAI) on day 1 of a 21 day cycle. Capecitabine starting dose of 500 mg/m2 by mouth twice daily, on days 1 - 14 of a 21 day cycle. Bevacizumab 10 mg/kg by vein on day 1 of a 21 day cycle.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab
- Oxaliplatin + Capecitabine (Experimental): Oxaliplatin 140 mg/m2 by Hepatic Arterial Catheter (HAI) on day 1 of a 21 day cycle. Capecitabine starting dose of 500 mg/m2 by mouth twice daily, on days 1 -14 of a 21 day cycle.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — 140 mg/m2 by Hepatic Arterial Catheter (HAI) on day 1 of a 21 day cycle.
  Other Names: Eloxatin
Drug: Capecitabine — Starting dose of 500 mg/m2 by mouth twice daily, on days 1 - 14 of a 21 day cycle.
  Other Names: Xeloda
Drug: Bevacizumab — 10 mg/kg by vein on day 1 of a 21 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: Oxaliplatin + Capecitabine + Bevacizumab

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of oxaliplatin and capecitabine with or without bevacizumab that can be given to patients with advanced cancer that has spread to the liver. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Oxaliplatin is designed to keep new cancer cells from growing.

Capecitabine is designed to interfere with the growth of cancer cells.

Bevacizumab is designed to block the growth of blood vessels that supply nutrients necessary for tumor growth. This may prevent or slow down the growth of cancer cells. Bevacizumab is no longer FDA approved to treat breast cancer.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study "arm" based on the results of your screening tests. All patients will receive oxaliplatin and capecitabine. If your doctor thinks it is in your best interest, you will also receive bevacizumab.

* If you are in Arm 1, you will receive oxaliplatin, capecitabine, and bevacizumab.
* If you are in Arm 2, you will receive oxaliplatin and capecitabine.

Arm 1:

You will be assigned to a dose level of capecitabine based on when you joined this study. Up to 4 dose levels of capecitabine will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of capecitabine is found.

All participants will receive the same dose levels of oxaliplatin and bevacizumab.

Arm 2:

You will be assigned to a dose level of capecitabine based on when you joined this study. Up to 4 dose levels of capecitabine will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of capecitabine is found.

All participants will receive the same dose levels of oxaliplatin.

Additionally, after the highest tolerable dose is found for each arm, if a certain tumor type is found to have responded well to the study drug combination, 14 participants with that tumor type will receive the study drugs at that dose level.

In each arm, after the highest tolerable dose of the study drug combination is found, up to 20 extra participants with any tumor type will receive that dose level.

Additionally, after the highest tolerable dose is found for each arm, if a certain tumor type is found to have responded well to the study drug combination, 14 participants with that tumor type will receive the study drugs at that dose level.

Catheter Placement for Study Drug Administration:

You will be hospitalized to receive the study drug combination. On the day of your admission to the hospital, you will have a catheter (a sterile flexible tube that will be placed in the hepatic artery [a blood vessel in the liver] while you are under local anesthesia) through which you will receive the study drugs. The catheter will be placed and removed during each cycle. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

You must lay in bed for the entire time that the catheter is in place. The catheter will either be removed right after your chemotherapy or it may remain in overnight.

Study Drug Administration:

Arm 1:

After completion of oxaliplatin and bevacizumab, you will receive a total of 28 doses of capecitabine, 1 dose twice daily. You will then receive bevacizumab by vein over 1½ hours. The first time you receive bevacizumab, it will be given over 90 minutes. If you tolerate it well, the rest of the doses will be given over 30-60 minutes.

On Days 1-14 of each cycle, you will take capecitabine by mouth 2 times each day. You should take it with a cup (8 ounces) of non-carbonated water within 30 minutes after a meal.

Arm 2:

On Day 1 of each 21-day cycle, you will receive oxaliplatin through the catheter over 2 hours.

After completion of oxaliplatin and bevacizumab, you will receive a total of 28 doses of capecitabine, 1 dose twice daily. You should take it with a cup (8 ounces) of non-carbonated water within 30 minutes after a meal.

Study Visits:

At each study visit, you will be asked about any other drugs you may be taking and about any side effects you may be having.

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn to test your blood's ability to clot.
* If you are able to become pregnant, you will have a urine pregnancy test.

At the end of every even cycle (Cycles 2, 4, 6, and so on):

* Blood (about 1 tablespoon) will be drawn to test for tumor markers.
* You will have scans to check the status of the disease. This may include a chest x-ray, CT scan, MRI scan, a PET scan, and/or a PET/CT scan. If the study doctor thinks it is more appropriate for you, other types of scans may need to be performed.

Length of Study:

You may continue taking the study drug combination for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug combination if the disease gets worse or intolerable side effects occur.

If the disease is only in your liver and you have responded to treatment, you may be eligible to receive surgery. If eligible, you will receive surgery 6 weeks after taking your last dose of study drugs if you are in Arm 1 or 4 weeks after taking your last dose of study drugs if you are in Arm 2. The study doctor will discuss this with you in more detail and you will sign a separate consent form if you have surgery.

Your participation on the study will be over once you have completed the follow-up visit.

Follow-Up Visit:

About 6 weeks after your last dose of study drugs, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a CT scan, MRI scan, PET scan, or PET/CT scan to check the status of the disease. If the study doctor thinks it is in your best interest, other types of scans may also be performed.

This is an investigational study. Oxaliplatin is FDA approved and commercially available for the treatment of colorectal cancer. Bevacizumab is FDA approved and commercially available for the treatment of colorectal and lung cancers. Capecitabine is FDA approved and commercially available for the treatment of colorectal and breast cancers.

Giving the study drugs together for advanced cancer is investigational.

Up to 116 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed cancer with predominant liver metastases.
2. Performance status Eastern Cooperative Oncology Group (ECOG) 0-2 (capable of all self care but unable to carry out any work activities).
3. Adequate renal function (creatinine clearance >50 mL/min).
4. Adequate liver function: total bilirubin </= 4 mg/dL, alanine transaminase (ALT) </= 5 times upper normal reference value. Patients with total bilirubin between 3.0 and 4.0 mg/dL must have blood ammonia level checked at baseline. Blood ammonia level must be within normal limits for enrollment.
5. Adequate bone marrow function (absolute neutrophil count (ANC) >/= 1000 cells/uL; platelets (PLT) >/= 70,000 cells/uL).
6. At least 3 weeks from prior cytotoxic chemotherapy or radiation therapy. If targeted or biologic therapy, there should be at least 5 half lives or 3 weeks, whichever is shorter, from day 1 of treatment.
7. All females in childbearing age MUST have a negative urine human chorionic gonadotropin (HCG) test before the first dose, unless prior hysterectomy or menopause (defined as age above 55 and six months without menstrual activity). Patients should not become pregnant or breast-feed while on this study. Sexually active patients should use effective birth control.
8. Ability and willingness to sign informed consent form.
9. Must be >/= 18 years of age.
10. Patients with unresectable liver-only (isolated liver) metastases are eligible; those who show adequate response may be considered for liver resection and/or radiofrequency ablation (RFA) of remaining disease.

Exclusion Criteria:

1. Pregnant females.
2. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
3. Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection requiring parental antibiotics, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patients already in uncompensated liver failure (i.e., Child Pugh Liver Classification C).
5. History of hypersensitivity to any component of the formulation.
6. Exclusion criteria only for patients enrolled in Arm 1: Serious or non-healing wound, ulcer, or bone fracture.
7. Exclusion criteria only for patients enrolled in Arm 1: Any history of abdominal fistula or gastrointestinal perforation; or intra-abdominal abscess within 28 days of enrollment.
8. Exclusion criteria only for patients enrolled in Arm 1: Uncontrolled systemic vascular hypertension (systolic blood pressure > 140 mm Hg, diastolic Blood Pressure > 90 mm Hg).
9. Exclusion criteria only for patients enrolled in Arm 1: History of bleeding CNS metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2010-09-30 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Hepatic Arterial IUnfusion (HAI) Oxaliplatin, with Oral Capecitabine, with or without Systemic Intravenous Bevacizumab | First 21 day cycle
  If more than 33% of patients enrolled in any particular dose level develop dose limiting toxicity (DLT), treatment will continue at dose level immediately below. If not more than 33% of the patients in cohort develop DLT, this cohort considered MTD. DLT defined as any grade 3 or 4 non-hematologic toxicity as defined in current version of NCI CTCAE, even if related to study medications (except nausea and vomiting, electrolyte imbalances responsive to appropriate regimens or alopecia), any grade 4 nausea or vomiting > 5 days despite maximum anti-nausea regimens, and any other grade 3 non-hematologic toxicity including symptoms/signs of vascular leak or cytokine release syndrome, but excluding alopecia; grade 4 thrombocytopenia; any grade 4 neutropenia of more than seven days duration, despite supportive care or associated with bleeding and/or sepsis; or any severe or life-threatening complication or abnormality not covered in NCI CTCAE. MTD defined by DLTs that occur in first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org